CLINICAL TRIAL: NCT04089514
Title: Pan-EU Real-World Experience With Imraldi®
Brief Title: A Real-world Study of Imraldi® Use
Acronym: PROPER
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: EUR-BIO-18-11391
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Arthritis, Rheumatoid (RA); Axial Spondyloarthritis (axSpA); Arthritis, Psoriatic (PsA); Crohn's Disease (CD); Colitis, Ulcerative (UC)
Keywords: Biologics; Non-interventional; Real-world; Adalimumab; Europe
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adalimumab Therapy: Adult participants diagnosed with immune-mediated inflammatory disease will receive adalimumab as a prescribed therapy
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Administered as specified in the treatment arm
  Other Names: Imraldi

SUMMARY:
The primary objective of this study is to evaluate candidate predictors of persistence on adalimumab (Imraldi®) participants diagnosed with immune-mediated inflammatory disease in Europe (EU).

The secondary objectives of this study are to describe participant clinical characteristics at baseline, utilization of Imraldi® over time, biologic drug effectiveness over time, participant satisfaction with biologic administration, routine laboratory values and clinical evaluation measurements over time, use of relevant concomitant medication use over time, immunogenicity of biosimilars and to summarize safety events.

ELIGIBILITY:
Inclusion Criteria:

* Initiation on Imraldi® therapy after 18th October 2018, as part of routine treatment immediately after transitioning from at least 16 weeks' treatment with originator adalimumab (Humira®)
* Availability of at least one Baseline disease score (i.e. within 16 weeks prior or up to 6 weeks post-initiation of Imraldi®)
* Should provide informed consent to participate in the study

Exclusion Criteria:

- Unlikely to attend for regular clinic visits for the duration of study follow-up, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with RA, or axSpA, or PsA, or CD, or UC, who are receiving biosimilar adalimumab (Imraldi®) therapy for their immune-mediated inflammatory disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Candidate Predictors of Persistence on Adalimumab | Baseline up to Week 48
  Candidate predictors (baseline clinical characteristics, disease score as applicable, incidence and clinical management of flares, and patient satisfaction survey) will be assessed via cox regression which will result in a hazard ratio.

SECONDARY OUTCOMES:
Number of Participants by Baseline Clinical Characteristic Categories | Baseline
  Baseline characteristics categories may include age, gender, diagnosis, duration of disease, relevant medical and surgical history, relevant co-morbidities, disease score, relevant concomitant therapies.
Number of Participants by Utilization of Adalimumab Categories | Baseline up to Week 48
  Adalimumab utilization categories may include type, dose, dose frequency and mode of administration, any changes, reason(s) for change and/or discontinuation.
Change from Baseline in Disease Scores as Applicable by Indication | Baseline up to Week 48
  Disease score as applicable by indication may include participant assessments of disease specific questionnaires (e.g. Disease Activity Score- 28 (DAS-28), Bath Ankylosing spondyloarthritis Functional Index (BASDAI), Harvey Bradshaw Index (HBI), Partial Mayo Score, Psoriatic Arthritis Response Criteria (PsARC))
Patient Satisfaction with Biologic Administration | Baseline up to Week 48
  Patient satisfaction with biologic administration will be assessed via a patient satisfaction questionnaire.
Number of Participants with Clinically Significant Laboratory Values and Clinical Evaluation Measurements | Baseline up to Week 48
  Clinical significance will be assessed by the investigator.
Number of Participants by Utilization of Relevant Concomitant Medication Categories | Baseline up to Week 48
  Concomitant medication utilization categories may include type, dose, and any changes in use of relevant concomitant therapy.
Number of Participants with Anti-drug Antibodies | Baseline up to Week 48
  Participants will be assessed for positive antibody results.
Number of Participants with Serious Adverse Events (SAEs) and Causally-related Non-serious Adverse Events (AEs) | Baseline up to Week 48
  An AE is any untoward medical occurrence that does not necessarily have a causal relationship with treatment. An SAE is any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (54):
- Belgium (9):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Herentals
  - Research Site, Kortrijk
  - Research Site, Liège
  - Research Site, Sijsele
  - Research Site, Turnhout
- Germany (16):
  - Research Site, Berlin
  - Research Site, Bruchhausen-Vilsen
  - Research Site, Burghausen
  - Research Site, Dresden
  - Research Site, Elmshorn
  - Research Site, Erfurt
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hamm
  - Research Site, Heidelberg
  - Research Site, Magdeburg
  - Research Site, Munich
  - Research Site, München
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Ratingen
- Research Site, Dublin, Ireland
- Italy (10):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Pavia
  - Research Site, San Giovanni Rotondo
  - Research Site, Siena
  - Research Site, Varese
- Spain (9):
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Donostia / San Sebastian
  - Research Site, Granada
  - Research Site, Mérida
  - Research Site, Sant Joan Despí
  - Research Site, Seville
  - Research Site, Terrassa
  - Research Site, Valladolid
- United Kingdom (9):
  - Research Site, Ashford
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Cambridge
  - Research Site, Kettering
  - Research Site, Luton
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Sussex

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Muller-Ladner U, Dignass A, Gaffney K, Jadon D, Matucci-Cerinic M, Lobaton T, Carron P, Gisbert JP, Pande I, Utzinger M, Addison J. The PROPER Study: A 48-Week, Pan-European, Real-World Study of Biosimilar SB5 Following Transition from Reference Adalimumab in Patients with Immune-Mediated Inflammatory Disease. BioDrugs. 2023 Nov;37(6):873-889. doi: 10.1007/s40259-023-00616-3. Epub 2023 Aug 26. PMID 37632666